CLINICAL TRIAL: NCT04253002
Title: Preventing Suicide in African American Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePaul University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LR060519PSY; 1R01MH1183182 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Suicide
Keywords: Suicide; African American Adolescents; Prevention; Coping; Hope; Hopelessness
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robinson's Culturally Adapted Coping with Stress Course (Experimental)
  Interventions: Behavioral: Robinson's Culturally Adapted Coping with Stress Course (A-CWS)
- Standard Care Control Condition (Active Comparator)
  Interventions: Behavioral: Standard Care Control Condition

INTERVENTIONS:
Behavioral: Robinson's Culturally Adapted Coping with Stress Course (A-CWS) — Participants randomized to the experimental condition will take part in the Adapted Coping with Stress Course (A-CWS). The A-CWS is a 15-session, cognitive-behavioral group intervention designed to develop and enhance African American youths' skills to adaptively cope with stress, using standard cognitive-behavioral strategies such as relaxation training and cognitive restructuring. Emphasis is given to the identification of individual and contextual factors associated with suicide risk and the unique day-to-day experiences of the youth, providing options for adaptive coping (e.g., positive thinking) that are culturally consistent. The A-CWS is structured and manualized to allow its transportability to service providers working in similar environments with similar youth.
  Arms: Robinson's Culturally Adapted Coping with Stress Course
Behavioral: Standard Care Control Condition — Students meeting criteria for study inclusion and randomized into the standard care condition will be referred to the school-based health center (SBHC) mental health provider for case management. Standard care may range from (1) brief intervention by the SBHC mental health provider to (2) outside referral to local community service providers; these determinations will be made by the SBHC mental health team.
  Arms: Standard Care Control Condition

SUMMARY:
The overarching aim of the Success Over Stress Prevention Project is to reduce African American youth suicide. This study examines the impact of a 15-session, group-delivered, culturally-grounded, cognitive-behavioral intervention (i.e., PI Robinson's Adapted-Coping with Stress Course [A-CWS]), on the outcomes of interest, when it is delivered by social workers who are indigenous to the school system. The main objectives of this project are to (a) determine whether the intervention is effective when facilitated by social workers who are indigenous to the school system and (b) enhance resilience, increase adaptive coping strategies, and reduce both intrapersonal and interpersonal violence among youth receiving the prevention intervention. It is expected that increases in adaptive coping will lead to an increased ability for youth to manage stressors, thereby decreasing the incidence of suicide and violence among the youth. In addition, it is expected that evidence of the intervention's effectiveness, when facilitated by social workers who are indigenous to the school system, will lead to greater dissemination and sustainability of the intervention, thus, providing access to effective intervention resources to greater numbers of African American youth.

DETAILED DESCRIPTION:
This study will establish the effectiveness of Robinson's Adapted-Coping with Stress Course (A-CWS) and test hypotheses pertaining to the mechanism of change by which the A-CWS reduces suicide risk. Additionally, this study is expected to augment current theoretical models of adolescent suicidality. This effectiveness trial will inform procedures for scaling up efficacious, high quality, and culturally-grounded suicide prevention programs for low-resourced, urban African American youth; as such, this study is practice relevant and expected to inform best practices for the prevention of suicide among African American adolescents. The specific aims are:

1. To examine the effectiveness of the A-CWS intervention, as delivered by social workers who are indigenous to the school system, to reduce active suicidal ideation, within a sample of low-resourced, urban African American adolescents.
2. To understand the mechanism by which the A-CWS intervention reduces suicide risk for low-resourced, urban African American adolescents.
3. To establish the fidelity of an evidence-based, culturally-grounded coping with stress intervention (i.e., the A-CWS), developed for low-resourced, urban African American adolescents, delivered by social workers indigenous to the school system.
4. To understand the extent that thwarted belongingness, perceived burdensomeness, and socio-ecological factors influence the development of active suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Students: Enrolled 9th grade student at time of initial enrollment at participating high school
* Parents/guardians: Child enrolled in study
* Teachers: Student enrolled in study

Exclusion Criteria:

* Not a 9th grade student at time of initial enrollment
* No parent/legal guardian permission
* For parents and teachers: no students enrolled in study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Suicide Ideation | Assessments will be administered through study completion, an average of every six months.
  Suicide ideation will be measured using the Suicidal Ideation Questionnaire (SIQ-JR), a 15-item measure of adolescents' distress and suicidal intent. Scale scores range from 0 to 90, with higher scores meaning a worse outcome (i.e., greater suicide ideation).

SECONDARY OUTCOMES:
Change in Adaptive Coping | Assessments will be administered through study completion, an average of every six months.
  Adaptive Coping will be measured using The Adolescent Coping Orientation for Problem Behaviors (A-COPE), which is a 54 item self-report questionnaire that measures coping strategies among adolescents
Change in Hope | Assessments will be administered through study completion, an average of every six months.
  Hope will be measured using the The Children's Hope Scale (CHS), a six-item self-report measure of children's perceived interpersonal competencies, including the belief that their goals can be met.
Change in Hopelessness | Assessments will be administered through study completion, an average of every six months.
  Hopelessness will be measured using the Hopelessness Scale for Children (HSC). The HSC consists of 17 true-false items. The domains measured include: feelings about the future, loss of motivation, and future expectations

CONTACTS AND LOCATIONS:
Overall Officials: LaVome Robinson, PhD, Principal Investigator — DePaul University
Locations (6):
- United States (6):
  - Richard T. Crane High School, Chicago, Illinois
  - DePaul University, Chicago, Illinois
  - Dunbar Vocational Career Academy, Chicago, Illinois
  - Orr Academy High School, Chicago, Illinois
  - Wendell Phillips Academy High School, Chicago, Illinois
  - Proviso East High School, Maywood, Illinois